CLINICAL TRIAL: NCT06128785
Title: Electroacupuncture Promotes Gastrointestinal Functional Recovery After Radical Colorectal Cancer Surgery: a Multicenter Randomized Controlled Study
Brief Title: Electroacupuncture (EA) Promotes Gastrointestinal Functional Recovery After Radical Colorectal Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: ShuGuang Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Baoshan hospital of Integrated Traditional Chinese and Western Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-144
Record Dates: First submitted 2023-09-04; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Gastrointestinal Dysfunction
Keywords: Colorectal Cancer; Gastrointestinal Dysfunction; Enhanced Recovery After Surgery; Electroacupuncture; Randomized Controlled Trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Needles: Huatuo brand disposable acupuncture needles φ0.25×40mm (1.5 inch); needles are purchased from Suzhou Medical Supplies Factory Co.
  Acupoint: bilateral Hegu (LI4), Zhigou (SJ6), Zusanli (ST36), Shangjuxu (ST37), lasting 30 min each time.
  Postoperative electroacupuncture stimulation method: all acupoints will be taken by tonifying method after obtaining qi, and unilaterally connected to the electroacupuncture instrument for electrical stimulation with a continuous wave frequency of 5 Hz and a stimulation intensity as tolerated by the patient for 30 min each time. Acupuncture stimulation will be given every 12 h. The duration of treatment was from postoperative to the fourth postoperative day (d0-d4) or until the patient's first postoperative anal discharge or until the fourth day.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both groups will use adhesive pads, and the sham acupuncture needle will have the same appearance as the traditional needle, with a blunt tip (Suzhou Medical Supplies Factory, specification 0.25×40mm), lifting and inserting and twisting, but not piercing the adhesive pad. The output wire of the special sham electroacupuncture apparatus is cut in the middle, and the appearance is as usual; that is, the electroacupuncture apparatus shows an on state, but is not actually energized; the electroacupuncture points, acupuncture time points, frequency, retention time, and duration of treatment are the same as the intervention group.
  All study patients will be treated independently and separately, ensuring that patients will not come into contact with each other. To test the effectiveness of blinding of participants, two hospitals will be selected from for blinded success assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Electroacupuncture group (Experimental): The acupuncture will be performed within 6 hours after surgery Acupoint: bilateral Hegu (LI4), Zhigou (SJ6), Zusanli (ST36), Shangjuxu (ST37), All acupoints will be taken by tonifying method after obtaining qi, and unilaterally connected to an electroacupuncture instrument for electrical stimulation with a continuous wave frequency of 5 Hz and a stimulation intensity as tolerated by the patient for 30 min each time. Acupuncture stimulation was given every 12 h. The duration of treatment was from postoperative to the fourth postoperative day (d0-d4) or until the patient's first postoperative anal discharge or until the fourth day.
  Interventions: Device: Electroacupuncture group
- Sham EA group (Sham Comparator): In order to achieve maximum patient blindness, both groups will use adhesive pads, and the sham acupuncture needle will have the same appearance as the traditional needle, with a blunt tip (Suzhou Medical Supplies Factory, specification 0.25×40mm), lifting and inserting and twisting, but not piercing the adhesive pad. The output wire of the special sham electroacupuncture apparatus is cut in the middle, and the appearance is as usual; that is, the electroacupuncture apparatus shows an on state, but is not actually energized; the electroacupuncture points, acupuncture time points, frequency, retention time, and duration of treatment are the same as the intervention group, and the patients are informed that it is an effective light current input and may not feel stimulation, but the current is output. All study patients will be treated independently and separately to ensure that patients will not come into contact with each other.
  Interventions: Other: Sham EA group
- Conventional control group (No Intervention): Routine perioperative management will be given, postoperative fluid and nutritional support, correction of acid-base imbalance, electrolyte disorders, anti-infection, hemostasis and other symptomatic management.

INTERVENTIONS:
Device: Electroacupuncture group — Acupoint: bilateral Hegu (LI4), Zhigou (SJ6), Zusanli (ST36), Shangjuxu (ST37). All acupoints will be taken by tonifying method after obtaining qi, and unilaterally connected to an electroacupuncture instrument for electrical stimulation with a continuous wave frequency of 5 Hz and a stimulation intensity as tolerated by the patient for 30 min each time. Acupuncture stimulation was given every 12 h. The duration of treatment was from postoperative to the fourth postoperative day (d0-d4) or until the patient's first postoperative anal exhaust or until the fourth day.
  Other Names: experimental group
  Arms: Electroacupuncture group
Other: Sham EA group — Sham acupuncture needle will have the same appearance as the traditional needle, with a blunt tip (Suzhou Medical Supplies Factory, specification 0.25×40mm), lifting and inserting and twisting, but not piercing the adhesive pad. The output wire of the special sham electroacupuncture apparatus is cut in the middle, and the appearance is as usual; that is, the electroacupuncture apparatus shows an on state, but is not actually energized; the electroacupuncture points, acupuncture time points, frequency, retention time, and duration of treatment are the same as the intervention group, and the patients are informed that it is an effective light current input and may not feel stimulation, but the current is output.
  Arms: Sham EA group

SUMMARY:
The goal of this clinical trial is to verify the efficacy of electroacupuncture in accelerating the recovery of gastrointestinal function after colorectal cancer surgery. The main questions it aims to answer are:

* Whether electroacupuncture can accelerate the recovery of gastrointestinal function in patients after colorectal cancer surgery.
* Whether electroacupuncture intervention is safe for postoperative colorectal cancer patients.

Participants will be randomized into 3 groups:

The conventional control group will receive postoperative rehydration and nutritional support, correction of acid-base imbalance and electrolyte disturbance, anti-infection, hemostasis and other symptomatic treatments.

In the electroacupuncture group, acupuncture will be performed within 6 hours after surgery on the basis of the conventional control group. Acupoint: bilateral Hegu (LI4), Zhigou (SJ6), Zusanli (ST36), Shangjuxu (ST37). Both after obtaining Qi, and unilaterally connected to the electroacupuncture instrument for electrical stimulation, the current frequency is continuous wave 5 Hz, the intensity of stimulation was as the patient tolerated, each time lasting 30 min. Acupuncture stimulation was given every 12 h. The course of treatment was terminated postoperatively until the fourth postoperative day (d0-d4) or until the patient showed the first postoperative anal exhaust or continued until the fourth day.

The sham acupuncture group will based on the conventional control group, using a blunt-tipped needle tip that do not pierce the adhesive pad.

DETAILED DESCRIPTION:
Colorectal cancer is the most common and predominant malignancy, and radical resection surgery, as the main method of current treatment for colon and gastrointestinal cancers, is performed on a large number of patients each year. Clinically, abdominal surgery causes the highest frequency of gastrointestinal dysfunction and the longest relative duration of dysfunction. A condition in which gastrointestinal function has not fully recovered after abdominal surgery is called gastrointestinal dysfunction. The common symptoms of postoperative gastrointestinal dysmotility are abdominal distension, abdominal pain, nausea and vomiting, diminished or even absent bowel sounds, loss of anal discharge, loss of bowel movements, and even secondary symptoms such as fever and pulmonary infection. It will adversely affect patients' postoperative quality of life to varying degrees, weaken their gastrointestinal barrier capacity, and severe gastrointestinal dysfunction can lead to complications such as electrolyte disorders, intestinal adhesions, intestinal obstruction, anastomotic fistula, and abdominal wall incision dehiscence in patients, as well as increase the social burden and the economic burden of patients. Some clinical reports show that acupuncture has good efficacy on gastrointestinal dysfunction, and acupuncture has effects on the gastrointestinal tract such as promoting gastrointestinal motility and reducing the inflammatory response of the gastrointestinal tract. In this study, a multicenter, randomized, blinded, sham acupuncture-controlled clinical design will be used to verify the efficacy of postoperative electroacupuncture in accelerating the recovery of gastrointestinal function after colorectal cancer surgery.

Participants will be randomized into 3 groups:

The conventional control group will receive postoperative rehydration and nutritional support, correction of acid-base imbalance and electrolyte disturbance, anti-infection, hemostasis and other symptomatic treatments.

In the electroacupuncture group, acupuncture will be performed within 6 hours after surgery on the basis of the conventional control group. Acupoint: bilateral Hegu (LI4), Zhigou (SJ6), Zusanli (ST36), Shangjuxu (ST37). Both after obtaining Qi, and unilaterally connected to the electroacupuncture instrument for electrical stimulation, the current frequency is continuous wave 5 Hz, the intensity of stimulation was as the patient tolerated, each time lasting 30 min. Acupuncture stimulation was given every 12 h. The course of treatment was terminated postoperatively until the fourth postoperative day (d0-d4) or until the patient showed the first postoperative anal exhaust or continued until the fourth day.

The sham acupuncture group will based on the conventional control group, using a blunt-tipped needle tip that do not pierce the adhesive pad. In other words, the electroacupuncture instrument show the state of being connected, but it is not actually energized; the acupuncture points, acupuncture time points, frequency, retention time and treatment duration were the same as those of the intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical patients who meet the diagnostic criteria for colorectal cancer and require elective radical colorectal cancer surgery;
2. 18 years old ≤ age ≤ 79 years old, with no restriction on gender;
3. Understand, agree to participate in this study and sign the informed consent form;
4. American society of Aneshesiologists (ASA) classification I to III.

Exclusion Criteria:

1. Patients with psychiatric disorders;
2. Patients who have participated or are participating in other clinical studies in the 3 months prior to enrollment;
3. Patients with severe malnutrition (NRS2002 score ≥ 3);
4. Patients with total colectomy;
5. Patients undergoing ileal diversion for rectal cancer;
6. Patients with tumor infiltration requiring resection of other organs;
7. Prophylactic fistulae.

Anyone who meets any of the above criteria will be excluded from the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-06 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Time of first postoperative exhaust | up to 4 days after surgery.
  The time between the patient's first exhaust and the end of surgery will be recorded.

SECONDARY OUTCOMES:
Time of first postoperative defecation | up to 4 days after surgery.
  Patients self-report their defecation and doctors record the time.
Length of recovery of bowel sounds after surgery ( Yueyang Hospital records only) | up to 4 days after surgery.
  Monitoring by continuous auscultation recorder of bowel sounds immediately at the end of surgery; Determination of recovery of postoperative bowel sounds: the time point when regular bowel sounds are observed and greater than 4 times/minute, calculate its time until the end of surgery (h), this outcome is only used in our center.
Time of first postoperative intake of water | up to 4 days after surgery.
  The time when the patient first entered water after surgery was recorded separately.
Number of Postoperative nausea and vomiting episods | up to 4 days after surgery.
  During the postoperative hospitalization, whenever nausea, vomiting and abdominal distension occur, patients or their family members use the uniform tabulation to record the occurrence time by themselves and inform the medical staff in time, and the medical staff keep records at the same time. The time until the end of the operation and the number of postoperative episodes will be calculated before discharge.
Quality of life scale 1 | baseline, discharge 1 day, 1 month after surgery.
  Version 3.0 European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), standard score, range from 0 to 100, higher scores mean a better outcome.
Quality of life scale 2 | baseline, discharge 1 day, 1 month after surgery.
  Short Form 12 scale (Chinese version). (Short Form 12 scale consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability).
Visual Analog Scale (VAS) of Pain | up to 4 days after surgery.
  Visual analogy score (0 to 5, higher scores mean a worse outcome)
Postoperative hospitalization days | up to 4 days
  Calculate and record the number of days from the day of surgery to the day of patient discharge.
Biochemical indexes 1 | 1 hour postoperatively, 12 hours postoperatively, 72 hours postoperatively.
  Hypersensitive C-reactiveprotein (hs-CRP), μg/L.
Biochemical indexes 2 | 1 hour postoperatively, 12 hours postoperatively, 72 hours postoperatively.
  Interleukin-6 (IL-6), μg/L.
Biochemical indexes 3 | baseline, discharge 1 day.
  serum albumin (ALB), g/L.

OTHER OUTCOMES:
Adverse Event Assessment | up to 4 days
  Any adverse events in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, M.D., Principal Investigator — Shanghai Yueyang Integrated Medicine Hospital
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting 12 months after publication.
Access Criteria: For academic communication only, online supplementary documents and email communication can be added.

REFERENCES:
- [Derived] Sun L, Wei X, Feng T, Gu Q, Li J, Wang K, Zhou J. Electroacupuncture promotes gastrointestinal functional recovery after radical colorectal cancer surgery: a protocol of multicenter randomized controlled trial (CORRECT trial). Int J Colorectal Dis. 2024 Dec 9;39(1):198. doi: 10.1007/s00384-024-04768-8. PMID 39652211